CLINICAL TRIAL: NCT04481100
Title: Phase II Study of Concurrent Chemoradiotherapy With Itraconazole in Treating Patients With Locally Advanced Esophageal Squamous Cancer
Brief Title: CCRT With Itraconazole in Locally Advanced Squamous Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shixiu Wu, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200707
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Esophageal Neoplasm; Esophageal Diseases; Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Concurrent chemoradiotherapy; Itraconazole; Hedgehog pathway
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases; Esophageal Squamous Cell Carcinoma | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): Itraconazole capsule 100mg twice daily for 6 weeks concurrent with chemoradation.
  Interventions: Drug: itraconazole

INTERVENTIONS:
Drug: itraconazole — Oral administration of itraconazole twice daily concurrent with chemoradiation

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of concurrent chemoradiotherapy combined with Itraconazole in patients with locally adcvanced esophageal squamous cancer

DETAILED DESCRIPTION:
Esophageal cancer is one of the most lethal malignancies. Esophageal squamous cell carcinoma (ESCC) is the predominant type in China, accounting for over 90% of all esophageal cancer. Concurrent chemoradiation therapy (CCRT) remains the standard therapy of locally advanced ESCC. However, the outcome remains poor.

The aberrant activation of Hedgehog (HH) signaling is associated with a variety of human malignancies. Previous studies found that the reactivation of HH pathway occurs in 60% of esophageal cancer. Targeting the Hh pathway for cancer therapy was expected to work wonders in Hh-dependent cancers. Itraconazole, an antifungal agent, has been shown to inhibit the Hh and AKT signaling pathways.

The aim of our study is to evaluate the efficacy and safety of concurrent chemoradiotherapy combined with Itraconazole in patients with locally adcvanced esophageal squamous cancer

ELIGIBILITY:
Inclusion Criteria:

age:18-75 years, male or femal.

Histologically or cytologically confirmed Squamous Cell Carcinoma of the Esophagus, locally advanced, unresectable disease.

Clinical staged T3-4N0M0, T1-4N+M0,Ⅱ-Ⅳa(AJCC 8th)

Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.

ECOG 0-1.

Adequate organ function.

Patient has given written informed consent.

Exclusion Criteria:

Unwilling or unable to provide informed consent

Known allergy to itraconazole

Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.

Complete obstruction of the esophagus, or patients who have the potential to develop perforation, or unable to swallow Itraconazole.

Other malignancy within 5 years prior to entry into the study, expect for curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers.

Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent.

Pregnancy or breast-feeding.

Decision of unsuitableness by principal investigator or physician-in-charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 4-8 weeks
  ORR was evaluated 4-8 weeks after completion of RT and was recorded according to RECIST, version 1.1

SECONDARY OUTCOMES:
Treatment-emergent adverse events | year 0 - year 1
  Incidence of treatment-emergent adverse events would be assessed based on the common toxicity criteria for adverse events version 4.0 (CTCAE v4.0) and EORTC criterion.
Local-regional free survival (LRFS) | year 0 - year 3
  LRFS was calculated from the date of treatment initiation to the date of documented failure.
Overall survival (OS) | year 0 - year 3
  OS was determined as the time (in months) between the first day of therapy and the last follow-up or the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital & Shenzhen Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No